CLINICAL TRIAL: NCT07378449
Title: The Effect of Hand Exercise Hoops on Labour Pain: A Randomized Controlled Single-Blind Study
Brief Title: The Effect of Hand Exercise Hoops on Labour Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Dogan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2025/727
Record Dates: First submitted 2026-01-18; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Labour Pain; Midwifery
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand Exercise Hoop Group (Experimental)
  Interventions: Device: Hand Exercise Hoop
- Control Group (No Intervention)

INTERVENTIONS:
Device: Hand Exercise Hoop — Participants assigned to the intervention group will use a soft hand exercise hoop in combination with guided breathing exercises during the active phase of labor. The intervention will begin at 4-5 cm cervical dilation and continue throughout the active phase. During each uterine contraction, participants will be instructed to inhale deeply at the onset of the contraction and to squeeze the hand exercise hoop while slowly exhaling as the contraction intensifies. As the contraction subsides, participants will release the hoop and return to normal breathing. The hand exercise hoop will be used continuously during contractions as a mechanical distraction and sensory stimulus. The intervention aims to reduce pain perception through activation of the gate control mechanism, distraction from pain stimuli, increased endorphin release, and regulation of the autonomic nervous system via controlled breathing. Participants will receive verbal guidance and support from healthcare staff throughout
  Arms: Hand Exercise Hoop Group

SUMMARY:
This randomized, single-blind controlled trial aims to evaluate the effect of using a hand exercise ring combined with breathing exercises on labor pain, anxiety, and childbirth satisfaction in primiparous women during the active phase of labor. Labor pain is a complex, multidimensional experience that intensifies as labor progresses and may lead to adverse physiological, psychological, and emotional consequences for both the mother and the fetus if not effectively managed. While pharmacological pain relief methods are effective, they may be associated with maternal and neonatal side effects and are not always accessible. Therefore, safe, low-cost, and non-pharmacological pain management strategies are of growing interest in maternity care.

The study will be conducted in a hospital labor ward and will include low-risk primiparous women aged 18-35 years who are admitted for vaginal birth. A total of 86 participants will be randomly assigned to either an intervention group or a control group. Women in the intervention group will receive a soft hand exercise ring and will be instructed to use it in conjunction with guided breathing exercises during uterine contractions, starting at 4-5 cm cervical dilation and continuing throughout the active phase of labor. During each contraction, participants will squeeze the hand exercise ring while exhaling and release it during relaxation periods between contractions. This intervention is designed to reduce pain perception through distraction, activation of the gate control mechanism, increased endorphin release, and regulation of the autonomic nervous system via controlled breathing.

The control group will receive routine intrapartum care without any additional pain management intervention. Outcome measures include labor pain intensity assessed using the Visual Analog Scale (VAS), anxiety levels measured with the State Anxiety Inventory (STAI Form TX-1), and childbirth satisfaction evaluated using the Maternal Satisfaction with Childbirth Scale. Pain and anxiety will be assessed at three stages of cervical dilation (4-5 cm, 6-7 cm, and 8-9 cm), while childbirth satisfaction will be assessed six hours postpartum.

The findings of this study are expected to contribute evidence regarding the effectiveness of a simple, non-invasive, and easily applicable intervention for labor pain management, potentially supporting its integration into routine midwifery care to improve women's childbirth experiences.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women with low-risk pregnancies

Exclusion Criteria:

* Women with high-risk pregnancies (such as preeclampsia, placenta previa)
* Women who will use any pharmacological or non-pharmacological pain management method
* Women who cannot be contacted or who are not amenable to referral

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2026-05-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Labor Pain Intensity | During the active phase of labor at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilation (up to 24 hours)
  Labor pain intensity will be assessed using the Visual Analog Scale (VAS), a validated tool consisting of a 10-cm horizontal line ranging from "no pain" (0) to "worst imaginable pain" (10). Participants will indicate their perceived pain intensity at each assessment point, with higher scores indicating greater pain severity.
Maternal Anxiety During Labor | During the active phase of labor at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilation (up to 24 hours)
  Maternal anxiety levels will be measured using the State Anxiety Inventory, a 20-item self-report questionnaire assessing situational anxiety. Total scores range from 20 to 80, with higher scores indicating higher levels of anxiety.
Maternal Satisfaction with Childbirth | Within 6 hours after vaginal birth.
  Maternal satisfaction with the childbirth experience will be evaluated using the Maternal Satisfaction with Childbirth Scale, a validated instrument assessing women's satisfaction with various aspects of the childbirth process. This study will use the vaginal birth version, which contains 43 items and 10 subscales to assess maternal satisfaction during childbirth. The subscales evaluate different areas of satisfaction related to the birth process (e.g., pain management, communication with healthcare personnel, birth environment). The total score range is 43-215. Higher total scores indicate greater satisfaction with the birth experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided